CLINICAL TRIAL: NCT01368731
Title: Prophylactic Endoscopic Coagulation for the Prevention of Bleeding in Endoscopic Mucosal Resection (EMR) of Large Sessile Colonic Polyps: A Multi-centre, Randomised Control Trial
Brief Title: Prophylactic Coagulation for the Prevention of Bleeding in Endoscopic Mucosal Resection of Large Sessile Colonic Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Dr Michael Bourke, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EMR-001-PEC; HREC2010/11/4.12(3155) AU RED (Other: HREC Office)
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Adenomatous Polyp of Large Intestine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- nil prophylactic coagulation (No Intervention)
- Prophylactic coagulation (Active Comparator)
  Interventions: Procedure: Prophylactic use of coagulation therapy

INTERVENTIONS:
Procedure: Prophylactic use of coagulation therapy — The procedure is completed as per usual, and if the patient has been randomized to the intervention group the appropriate coagulation therapy will be applied immediately after standard EMR to visible vessels within the mucosal resection area.
  Other Names: Heat probe; Soft coagulation
  Arms: Prophylactic coagulation

SUMMARY:
The hypothesis of this study is that prophylactic coagulation therapy with coagulation forceps to visible vessels within the mucosal defect for colonic Endoscopic Mucosal Resection (EMR) will reduce the rate of delayed bleeding when compared with current established standard EMR technique.

DETAILED DESCRIPTION:
Delayed bleeding from the site of the resection remains one of the most common complications following EMR, occurring in up to 12% of patients. The purpose of the study is to prevent such bleeding with the use of a technique known as: "coagulation therapy." This therapy involves using a small dose of heat energy that results in clotting(coagulation) of a blood vessel. It is already used widely in the stomach and we intend using this on a lower setting to blood vessels that are exposed after the resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to Westmead Hospital Endoscopy unit for endoscopic removal of a large sessile colonic polyp sized >20mm
* Age >18 years
* Able to give informed consent to involvement in trial

Exclusion Criteria:

* Pregnancy: currently pregnant or attempting to become pregnant
* Lactation: currently breastfeeding
* Taken clopidogrel within 7 days
* Taken warfarin within 5 days
* Had full therapeutic dose unfractionated heparin within 6 hours
* Had full therapeutic dose low molecular weight heparin (LMWH) within 12 hours
* Known clotting disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2011-05; Primary Completion 2014-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Presence of delayed bleeding | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, Principal Investigator — Westmead Hospital - Endoscopy Unit
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Bahin FF, Naidoo M, Williams SJ, Hourigan LF, Ormonde DG, Raftopoulos SC, Holt BA, Sonson R, Bourke MJ. Prophylactic endoscopic coagulation to prevent bleeding after wide-field endoscopic mucosal resection of large sessile colon polyps. Clin Gastroenterol Hepatol. 2015 Apr;13(4):724-30.e1-2. doi: 10.1016/j.cgh.2014.07.063. Epub 2014 Aug 20. PMID 25151254